CLINICAL TRIAL: NCT01125735
Title: A Prospective, Randomized, Controlled Study of MIST Therapy's Effectiveness in Wound Bed Preparation and the Role of Bacterial Biofilm in Subjects Presenting With Chronic, Non-healing Wounds
Brief Title: MIST Therapy's Effectiveness in Wound Bed Preparation and Role of Bacterial Biofilm in Chronic, Non-healing Wounds
Acronym: Celleration
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Contract negotiations were terminated and study never started.
Sponsor: Georgetown University (Other)
Collaborators: Celleration, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Chief of the Division of the Center for Wound Healing, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-093
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Nonhealing Wounds
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIST Therapy (Experimental): MIST Therapy is a low energy, low intensity ultrasound delivered through a saline mist to the wound bed.
  Interventions: Device: MIST Therapy
- Standard of Care (Other): Standard of Care with saline rinse using a sham device which is a nebulizer compressor designed to deliver a continuous saline mist to a skin treatment site. The saline mist generated has been designed to be comparable to that delivered by the MIST Therapy System, but without the ultrasound waves.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: MIST Therapy — The MIST Therapy System is designed to deliver therapeutic ultrasound to the wound bed without direct contact of the device to the body (noncontact). The system generates and propels the therapeutic MIST Therapy towards the tissue. The saline solution is directed to the tip surface and is atomized through the vibration of the tip surface. This surface creates atomization of the fluid, breaking it apart into small particles of uniform size. Once the particles of fluid are released from the tip, a second phenomenon, the acoustic pressure wave, drives them toward the wound.
  Arms: MIST Therapy
Other: Standard of Care — Standard of Care with saline rinse using a sham device which is a nebulizer compressor designed to deliver a continuous saline mist to a skin treatment site. The saline mist generated has been designed to be comparable to that delivered by the MIST Therapy System, but without the ultrasound waves.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of MIST Therapy in combination with standard of care (SOC) compared to SOC alone on reducing the bacteria in your wound and preparing the wound bed for surgical closure in patients that have chronic, non-healing wounds.

The MIST Therapy System delivers therapeutic ultrasound to the wound bed without direct contact. Saline solution is converted into fine particles and released towards the wound by sound pressure waves to remove dead or damaged tissue. The MIST Therapy System is currently the only FDA cleared non-contact ultrasound device to promote wound healing.

Standard of care procedures include surgical debridement of the wound in the operating room to remove all infected, dead tissue and bone.

This research is being done because the investigators do not know which of these commonly-used treatments is better, and because the investigators would like to evaluate the bacteria that is present in the wound.

DETAILED DESCRIPTION:
The trial is designed as an investigator-initiated prospective, randomized, controlled single blinded study, at a single study center, of persons presenting with a chronic, non-healing wound the knee with a potential for rapid deterioration, leading to limb loss. Chronic wounds defined as, having been present longer than 30 days and have failed to demonstrate greater than about a 50% reduction in surface area in the previous 30 days despite the administration of appropriate and standard wound care as well as cases presenting with acute gangrene or massive tissue loss that do not meet the 30 day criteria will be included. All wounds must be at least 5 cm2. A SOC Doppler assessment will be performed to ensure that the wound is adequately vascularized.

For subjects who present with multiple chronic, non-healing wounds, only the largest wound meeting the entrance criteria will be enrolled in the study. This will be referred to as the patient's "index wound." Once a wound is designated as the "index wound," that wound will remain the index wound for the duration of the patient's study participation.

Adult patients with ESRD and who have a chronic, non-healing wound consenting to the study will be screened for eligibility and if subjects meet all the inclusion and none of the exclusion criteria, they will be enrolled for study participation. Enrolled patients will then be randomized to receive one of two treatment courses: a) MIST Therapy in conjunction with Standard of Care (SOC) (treatment group) or, b) SOC only using a Sham device (control group). The Sham device is a nebulizer compressor designed to deliver a continuous saline mist to a MIST Therapy System, but without the ultrasound waves. Both groups will have a primary closure (ie. split thickness skin graft or delayed primary closure) as part of the eventual treatment plan. Both groups will undergo up to 5 SOC surgical debridements in the OR setting, with each debridement immediately followed by the subject's assigned study treatment.

Prior to initiating the assigned study treatment, a randomized patient will be required to undergo a Baseline Evaluation. The Baseline Evaluation will include: wound area measurement, wound bed evaluation, and digital photograph. Following the Baseline Evaluation, a study patient will undergo surgical debridement of the index wound in the operating room setting. During this time, a tissue sample will be obtained prior to debridement in both study groups. A second tissue sample will be obtained from both study groups immediately following debridement (either SOC debridement or MIST therapy, depending on which group the patient was randomized into). These tissue samples will be utilized to assess the presence of biofilm in the wound prior to and following the assigned study treatment. A tissue sample will be taken in the form of a 2mm punch biopsy that will be obtained from the center of the wound as well as the wound margin in both study groups prior to debridement and immediately following debridement (either SOC debridement or MIST therapy, depending on which group the patient was randomized into). Along with SOC wound cultures, a swab of the wound will be taken before and after the treatment at the first OR visit and be sent to the Georgetown University lab for quantitative analysis of the bacteria present.

Following the Baseline evaluation and surgical debridement, study subjects will undergo up to 4 subsequent Interim Study Evaluations. The Interim Study Evaluations will include a wound assessment, wound measurements, digital photographs, and an adverse event assessment, and will be conducted at a frequency determined appropriate by the Principal Investigator until the wound bed appears appropriate for primary closure. As part of each Interim Study Evaluation, study subjects will undergo a subsequent surgical debridement in the OR setting, immediately followed by the assigned study treatment, (i.e., sham device with saline rinse or MIST therapy). Prior to each subsequent surgical debridement, a SOC wound culture and quantitative wound culture will be obtained for analysis.

Final tissue biopsies, from the wound center and wound margin, will be obtained prior to the primary closure procedure. Following definitive wound closure procedure, split thickness skin graft or delayed primary wound closure, the subject will undergo Bi-Monthly Wound Assessment, being followed for a maximum of 20 weeks from the date of his/her first surgical debridement. A Bi-Monthly Wound Assessment will include an assessment of maintained wound closure and an adverse event assessment.

SOC post-operative dressings may include Moist Wound Therapy and the use of Negative Pressure Wound Therapy. NOTE: No impregnated dressings will be allowed during the study period. No topical antibiotics or antibiotic dressings, topical antiseptics (silver, iodine, etc.), or antimicrobials will be allowed. The use of EMLA Cream is not allowed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years or older.
* Subject has a chronic non healing wound located below the knee.
* Subject's wound is 5 cm2 or larger
* Subject's wound is adequately vascularized, demonstrated by SOC Doppler assessment.
* Subject must sign an institutional review board (IRB) approved informed consent.
* Subject is willing and able to complete required follow up.
* Subject's wound has been present longer than 30 days without 50% reduction in surface area in previous 30 days.

OR

* Subject's wound presents with acute gangrene or massive tissue loss that does not meet the 30 day criteria.

Exclusion Criteria:

* Subject's wound requires the use of topical antibiotics at the time of study enrollment.
* subject's wound presents with a malignancy in the wound bed.
* Subject has a cardiac pacemaker or other electronic device implants.
* Subject has a disorder or situation that the investigator believes will interfere with study compliance.
* Subject is currently enrolled or enrolled in the last 30 days in another investigational device or drug trial.
* Subject is pregnant or pregnancy is suspected.
* Subject's wound is smaller than 5cm2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Healing | 20 weeks
  To compare the rate of healing at 20 weeks between the MIST therapy group and the control group and to compare the clinical effectiveness between the treatment groups in achieving appropriate wound bed preparation for a delayed primary closure procedure.

SECONDARY OUTCOMES:
Role and Presence of biofilm | 20 weeks
  To evaluate the role and presence of biofilms in chronic wounds in persons with ESRD undergoing MIST therapy as compared to the control group and to evaluate if the presence of a biofilm is reflected in the quantitative wound culture

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, MD, Principal Investigator — Georgetown Hospital